CLINICAL TRIAL: NCT03353246
Title: Assessment of Accuracy, Precision, and Feasibility of a Handheld Near-Infrared Light Device (InfraScanner 2000™) in Detecting Subdural and Epidural Hematomas in Patients Admitted to Duke University Hospital: A Pilot Study
Brief Title: Assessment of InfraScanner 2000™ in Detecting Subdural and Epidural Hematomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00087011
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Results first posted 2019-05-28 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-04

CONDITIONS: Head Trauma; Craniocerebral Injuries; Crushing Skull Injury; Head Injuries; Head Injuries, Multiple; Head Injuries, Closed; Head Trauma,Closed; Head Trauma Injury; Head Trauma, Penetrating; Head Injury, Minor; Head Injury Major; Head Injury, Open; Injuries, Craniocerebral; Injuries, Head; Multiple Head Injury; Trauma, Head
MeSH Terms: conditions — Craniocerebral Trauma; Head Injuries, Closed; Head Injuries, Penetrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- InfraScanner 2000™ (Experimental): All patients entered onto the trial will undergo at least one cranial scanning using the InfraScanner 2000™ within 30 minutes of CT. Patients will be scanned using the InfraScanner 2000™ within 30 minutes of each subsequent CT. Patients will know the results of the CT but not the InfraScanner 2000™. The standard for comparison will be determined as follows. A CT result that is positive for hematoma will be considered a true positive and a CT result that is negative for hematoma will be considered a true negative. In cases where the results of the CT are negative for hematoma and the results of the InfraScanner 2000™ are positive consideration of further follow-up will be given on a case-by-case basis.
  Interventions: Device: InfraScanner 2000™

INTERVENTIONS:
Device: InfraScanner 2000™ — The Infrascanner is a portable screening device that uses Near-Infrared (NIR) technology to screen patients for intracranial bleeding, identifying those who would most benefit from immediate referral to a CT scan and neurosurgical intervention.

SUMMARY:
The goal of this study is to determine the sensitivity, specificity, and positive and negative predictive values of the a portable near-infrared-based device (portable NIR-based device), the InfraScanner 2000™, to detect intracranial hematomas (epidural hematomas (EDH) and/or subdural hematomas (SDH)) in patients hospitalized at Duke University Hospital (DUH) who have sustained or who are suspected to have sustained head trauma and have consequently received a brain computed tomography (CT) scan(s).

DETAILED DESCRIPTION:
When applicable (conscious patient and/or family or legally authorized representative is present) the study will be introduced to the patient and relevant parties prior to the research team approaching the patient. While head trauma frequently results in impaired cognition and/or consciousness, and due to the urgency of these circumstances patients are often not accompanied by kin, whenever appropriate, the purpose of the research and the procedure will be explained in detail with all questions answered to the patient's and/or representative's satisfaction. Because patients who sustain head trauma injuries typically remain within the hospital for multiple days for monitoring and care, each participant may undergo multiple CT scans over the course of his or her hospitalization, affording the opportunity to one to numerous measurements from each patient during his or her hospital stay.

Within 30 minutes following each CT scan, the study team will approach the patient to scan the patient's cranium with the InfraScanner 2000™ (Image A). The procedure will entail placing 8 plastic light guides upon the patient's scalp. The study team member will use the device to sequentially emit light through each of the 8 light guides so that the light is incident upon scalp (Image B). The device is engineered such that the light emitter and receiver are spaced ~4cm apart, allowing the light's intensity to be measured between adjacent light guides (Image C). This entire procedure, including greeting the patient, placing the light guides, gathering the data, and removing the light guides should take ~10 minutes each time. The number of CT scans the patient receives determines the number of potential data collections. The patient will be approached by the study team following each CT scan to be scanned with the InfraScanner 2000™ (20). The patient and/or representative may refuse a scan during any encounter, and as such, the scan will not be done. For each patient scanned with the InfraScanner 2000™ they will be de-identified with a subject number, with age, sex, gender, skin color, hair color, hair thickness, mechanism of injury, Glasgow Coma Scale score, and mean time elapsed between CT scan and near-infrared measurement. These data will be stored in de-identified form on Research Electronic Data Capture (REDCap) and/or Microsoft Excel 2016 on a secured DHTS server (S:\NSU_IRB\Pro00087011).

The collection period for each research subject concludes 30-days following his or her initial measurement with the InfraScanner 2000™, patient discharge, or patient death.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who presents to Duke University Hospital with suspected head trauma and receives a brain CT scan will be considered for this study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haglund, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | InfraScanner 2000™
Started | 500
Completed | 500
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (25.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211
  Male | 289
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 104
  Not Hispanic or Latino | 396
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 10
  Black or African American | 168
  White | 231
  More than one race | 63
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 500

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of InfraScanner 2000 TM to Detect Any Size Hematoma at the Patient Level
Description: Percentage of subjects with hematomas detected by CT who had hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: For participants who had more than one scan, the first scan was used.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
percentage | 85.6 [78.8 to 92.3]

2. Primary Outcome: Sensitivity of InfraScanner 2000 TM to Detect Any Size Hematoma at the Scan Level
Description: Percentage of CT scans with hematomas detected that had hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: Among 500 patients, 443 had only one measurement (CT and InfraScan), 37 had two measurements, 16 had three measurements, 4 had four measurements.
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: Scans
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
Number analyzed (Scans) | 581
percentage | 88.5 [83.8 to 93.1]

3. Primary Outcome: Specificity of InfraScanner 2000 TM for Detection of Any Size Hematoma at the Patient Level
Description: Percentage of patients with no hematomas detected by CT who had no hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: For participants who had more than one scan, the first scan was used.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
percentage | 95.7 [93.7 to 97.7]

4. Primary Outcome: Specificity of InfraScanner 2000 TM for Detection of Any Size Hematoma at the Scan Level
Description: Percentage of CT scans with no hematomas detected that had no hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: Scans
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
Number analyzed (Scans) | 581
percentage | 95.5 [93.5 to 97.5]

5. Primary Outcome: False Positive Rate of InfraScanner 2000 TM for Detection of Any Size Hematoma at the Patient Level
Description: Percentage of patients with no hematomas detected by CT that had hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: For participants who had more than one scan, the first scan was used.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
percentage | 16.0 [9.1 to 23.0]

6. Primary Outcome: False Positive Rate of InfraScanner 2000 TM for Detection of Any Size Hematoma at the Scan Level
Description: Percentage of scans with no hematomas detected by CT that had hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: Scans
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
Number analyzed (Scans) | 581
percentage | 10.1 [5.7 to 14.5]

7. Primary Outcome: False Negative Rate of InfraScanner 2000 TM for Detection of Any Size Hematoma at the Patient Level
Description: Percentage of patients with hematomas detected by CT that had no hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: For participants who had more than one scan, the first scan was used.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
percentage | 3.8 [1.9 to 5.7]

8. Primary Outcome: False Negative Rate of InfraScanner 2000 TM for Detection of Any Size Hematoma at the Scan Level
Description: Percentage of scans with hematomas detected by CT that had no hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: Scans
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 500
Number analyzed (Scans) | 581
percentage | 5.2 [3.1 to 7.4]

9. Secondary Outcome: Sensitivity in Identification of Hematomas Within Detection Limits, at the Patient Level
Description: Percentage of subjects with hematomas within detection limits detected by CT who had hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: For participants who had more than one scan, the first scan was used. Analysis was completed in a subset of participants who had hematomas within detection limits.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 482
percentage | 94.2 [89.2 to 99.1]

10. Secondary Outcome: Specificity in Identification of Hematomas Within Detection Limits, at the Patient Level
Description: Percentage of patients with no hematomas within detection limits detected by CT who had no hematoma detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 482
percentage | 95.7 [93.7 to 97.7]

11. Secondary Outcome: Sensitivity for Bleeds Within Detection Limits by Hematoma Type at the Patient Level
Description: Percentage of subjects with hematomas within detection limits detected by CT that were detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: Estimates by hematoma type are not mutually exclusive; patients with multiple hematoma types are included in more than one estimate.
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: Hematomas
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 482
Number analyzed (Hematomas) | 98
percentage
  epidural hematoma (EDH): number analyzed (Hematomas) | 6
  epidural hematoma (EDH) | 100.0 [54.1 to 100.0]
  subdural hematoma (SDH): number analyzed (Hematomas) | 64
  subdural hematoma (SDH) | 96.9 [92.6 to 100.0]
  subarachnoid (SAH): number analyzed (Hematomas) | 12
  subarachnoid (SAH) | 75.0 [50.5 to 99.5]
  intracerebral (IH): number analyzed (Hematomas) | 16
  intracerebral (IH) | 100.0 [79.4 to 100.0]

12. Secondary Outcome: False Negative Value for Bleeds Within Detection Limits by Hematoma Type at the Patient Level
Description: Percentage of subjects with hematomas within detection limits detected by CT where no hematoma was detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 482
percentage
  epidural hematoma (EDH): number analyzed (Participants) | 6
  epidural hematoma (EDH) | 0.0 [0.0 to 0.97]
  subdural hematoma (SDH): number analyzed (Participants) | 64
  subdural hematoma (SDH) | 0.5 [0.0 to 1.3]
  subarachnoid (SAH): number analyzed (Participants) | 12
  subarachnoid (SAH) | 0.8 [0.0 to 1.7]
  intracerebral (IH): number analyzed (Participants) | 16
  intracerebral (IH) | 0.0 [0.0 to 0.97]

13. Secondary Outcome: Sensitivity for Bleeds Within Detection Limits by Hematoma Type at the Scan Level
Description: Percentage of CT scans with hematomas within detection limits detected by CT that were detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: CT scans
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 482
Number analyzed (CT scans) | 180
percentage
  epidural hematoma (EDH): number analyzed (CT scans) | 10
  epidural hematoma (EDH) | 90.9 [73.9 to 100.0]
  subdural hematoma (SDH): number analyzed (CT scans) | 119
  subdural hematoma (SDH) | 98.3 [96.0 to 100.0]
  subarachnoid (SAH): number analyzed (CT scans) | 25
  subarachnoid (SAH) | 88.0 [75.3 to 100.0]
  intracerebral (IH): number analyzed (CT scans) | 26
  intracerebral (IH) | 96.2 [88.8 to 100.0]

14. Secondary Outcome: False Negative Value for Bleeds Within Detection Limits by Hematoma Type at the Scan Level
Description: Percentage of CT scans with hematomas within detection limits detected by CT where no hematoma was detected by Infrascanner 2000 TM.
Time Frame: Up to 30 days after first CT scan
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: CT scans
Arm/Group | InfraScanner 2000™
Number analyzed (Participants) | 482
Number analyzed (CT scans) | 180
percentage
  epidural hematoma (EDH): number analyzed (CT scans) | 10
  epidural hematoma (EDH) | 0.3 [0.0 to 0.8]
  subdural hematoma (SDH): number analyzed (CT scans) | 119
  subdural hematoma (SDH) | 0.5 [0.0 to 1.3]
  subarachnoid (SAH): number analyzed (CT scans) | 25
  subarachnoid (SAH) | 0.8 [0.0 to 1.7]
  intracerebral (IH): number analyzed (CT scans) | 26
  intracerebral (IH) | 0.3 [0.0 to 0.8]

ADVERSE EVENTS:
Time Frame: During the time of the scan with the InfraScanner, up to 10 minutes
Arm/Group | InfraScanner 2000™
All-Cause Mortality (participants affected / at risk) | 0/500
Serious Adverse Events (participants affected / at risk) | 0/500
Other Adverse Events (participants affected / at risk) | 0/500

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT03353246/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT03353246/SAP_001.pdf